CLINICAL TRIAL: NCT03980041
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Active-Control Study to Evaluate the Efficacy and Safety of Nivolumab Administered in Combination With IPI-549 Compared to Nivolumab Monotherapy in the Treatment of Patients With Immune Therapy-Naïve, Advanced Urothelial Carcinoma
Brief Title: Study to Evaluate the Efficacy/Safety of IPI-549 in Combination With Nivolumab in Patients With Advanced Urothelial Carcinoma (MARIO-275)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPI-549-02
Record Dates: First submitted 2019-04-22; First posted 2019-06-10 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Solid Tumor; Advanced Cancer
Keywords: eganelisib; IPI-549
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — IPI-549; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IPI-549 + Nivolumab (Experimental): Participants receive IPI-549 orally (PO) daily in combination with nivolumab IV infusion every 4 weeks
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Placebo + Nivolumab (Active Comparator): Participants receive placebo orally (PO) daily in combination with nivolumab IV infusion every 4 weeks
  Interventions: Drug: Nivolumab; Drug: Placebos

INTERVENTIONS:
Drug: IPI-549 (eganelisib) — IPI-549 (40mg QD) administered orally in 28-day cycles
  Other Names: IPI549
  Arms: IPI-549 + Nivolumab
Drug: Nivolumab — Nivolumab (480mg Q4W) administered intravenously (IV) in 28-day cycles
  Other Names: OPDIVO®
Drug: Placebos — Placebo administered orally in 28-day cycles
  Other Names: Placebo
  Arms: Placebo + Nivolumab

SUMMARY:
The purpose of this study is to measure the effect of IPI-549 in combination with nivolumab when compared to nivolumab monotherapy in advanced urothelial cancer patients.

DETAILED DESCRIPTION:
Study IPI-549-02 is a multi-national, prospective, randomized, active-control Phase II trial to evaluate the efficacy and safety of IPI 549 administered in combination with nivolumab compared to nivolumab monotherapy.

The study will enroll approximately 160 checkpoint-naïve, advanced urothelial cancer patients who have progressed or recurred following treatment with platinum-based chemotherapy. Patients will be randomized 2:1 to receive intravenous (IV) nivolumab 480 mg every 4 weeks (Q4W) in combination with oral (PO) IPI 549 40 mg once daily (QD) or IV nivolumab 480 mg Q4W in combination with placebo PO QD.

Eligible patients who have confirmed progression of disease during treatment with nivolumab monotherapy may crossover to the combination treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra
* Measurable disease by CT or MRI as defined by RECIST v1.1
* Disease progression or recurrence after treatment:
* i) With at least 1 platinum-based chemotherapy regimen for the treatment of metastatic (Stage IV) or locally advanced unresectable disease; or
* ii) With disease recurrence within 1 year of completing a platinum-based neoadjuvant or adjuvant therapy
* Subject that have received more than 2 prior lines of chemotherapy must not have liver metastases
* Tumor tissues (archived or new biopsy) must be provided for biomarker analysis
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Blood sample must be provided for mMDSC levels for randomization into the study

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Any serious or uncontrolled medical disorder that may interfere with study treatment/interpretation
* Prior malignancy active within the previous 3 years except for local or organ confined early stage cancer that has been apparently cured
* Active, known, or suspected autoimmune disease
* A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 day of study drug administration
* Prior therapy with anti-tumor vaccines, any T cell co-stimulation or checkpoint pathways, or IPI-549
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption
* Past medical history of interstitial lung disease
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control
* Positive test for hepatitis B, C or HIV
* Dependent on continuous supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECISTv1.1 | First dosing date to date of confirmed disease progression, assessed up to 24 months
  ORR is defined as best response of complete response (CR) or partial response (PR) as measured by RECIST v1.1.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors. CR= Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.

SECONDARY OUTCOMES:
Time to Response (TTR) | First dosing date to date of first objective response, assessed up to 24 months
  TTR is defined as the time from the first dose of study treatment to first objective response [complete response (CR) or partial response (PR)] in patients with CR or PR.
Duration of Response (DOR) | Date of first objective response to date of confirmed disease progression, assessed up to 24 months
  DOR is defined as the time from the first objective response (CR or PR) to documented disease progression in patients with CR or PR.
Progression-Free Survival (PFS) | First dosing to date to confirmed disease progression or death, assessed up to 48 months
  PFS is defined as the time from the first dose of study treatment to documented disease progression or death due to any cause.
Changes from baseline in thyroid stimulating hormone (TSH) | Pre-treatment (within 7 days of first dose) to date of confirmed disease progression, assessed up to 24 months
  If TSH result is abnormal, subsequent testing of Free T3 and free T4 required.
Changes from baseline in electrocardiograms (ECGs) | Screening to date of confirmed disease progression, assessed up to 24 months
  ECGs assess heart problems by measuring the electrical activity generated by the heart as it contracts. The components that will be assessed during the ECG are P wave, QRS complex, ST segment, and T wave.
Changes from baseline in Eastern Cooperative Oncology Group (ECOG) performance | Screening to date of confirmed disease progression, assessed up to 24 months
  ECOG performance status describes the level of impact that disease has on the patient's daily living abilities. Scale ranges from 0 (Fully active and able to carry on all pre-disease performance without restriction) to 5 (Dead).
Population Pharmacokinetics (PK) of IPI-549-01 | Pre-dose, 0.5, 1.5, 3 and 6 hours following administration on Day 1 of Cycles 1 and 2 (each cycle is 28 days)
  IPI-549 blood concentrations in ng/mL.
Pharmacokinetics (PK) of Nivolumab | Pre-infusion and within 2 minutes of end of infusion on Day 1 of Cycles 1 and 4; Pre-infusion on Day 1 of Cycles 2 and 3, and every 4 cycles starting at Cycle 5 (each cycle is 28 days)
  Nivolumab blood concentrations will be assayed in ug/mL.
Changes from baseline in pulse rate | Screening to date of confirmed disease progression, assessed up to 24 months
  Pulse rate as measured in beats per minute (bpm)
Changes from baseline in temperature | Screening to date of confirmed disease progression, assessed up to 24 months
  Temperature as measured in celsius.
Changes from baseline in respiration rate | Screening to date of confirmed disease progression, assessed up to 24 months
  Respiration rate as measured in breaths per minute.
Changes from baseline in blood pressure | Screening to date of confirmed disease progression, assessed up to 24 months
  Systolic and diastolic blood pressure as measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Halle Zhang, PhD, RN, Study Director — Infinity Pharmaceuticals, Inc.
Locations (29):
- United States (7):
  - Parkview Physicians, Fort Wayne, Indiana
  - University of MD - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Center, Detroit, Michigan
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Bon Secours St. Francis Cancer Center, Greenville, South Carolina
  - Sarah Cannon Tennessee Oncology, Nashville, Tennessee
- Onkologicka Klinika, Prague, Czechia
- France (5):
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
- Italy (3):
  - Istituto per la Ricerca e la Cura del Cancro (IRCC), Candiolo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Nazionale dei Tumori, Napoli
- Poland (3):
  - Oddzial Chorob Rozrostowych Wojewodzki Szpital, Lodz
  - Dzienny Oddzial Chemioterapii, Racibórz
  - EXAMEN sp, Skorzewo
- Serbia (2):
  - Clinical Centre of Serbia, Belgrade
  - Institute for Oncology of Vojvodina, Kamenitz
- Spain (8):
  - ICO Institute Catalan of Oncology, Barcelona
  - Hospital de Sant Creu i Sant Pau, Barcelona
  - IMQ Zorrotzaurre, Bilbao
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitatio HM Sanchinarro, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.infi.com/home/our-development-program/ipi-549/